CLINICAL TRIAL: NCT02300831
Title: LUMINIST: LUng Cancer Molecular Insights Non Interventional Study
Acronym: LUMINIST
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: D1532R00004
Record Dates: First submitted 2014-11-18; First posted 2014-11-25 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: NSCLC
Keywords: NSCLC; Lung Cancer; SELECT-1; SELECT-2; selumetinib; biomarker; NIS; Observational study; Disease registry; Clinical Outcomes
MeSH Terms: conditions — Lung Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — All samples used in the study are collected under the auspices of the SELECT 1 study screening. Luminist provides the clinical data to correlate the with sample results.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NSCLC: The eligible patient population of this study will comprise of advanced 2nd line NSCLC patients who are screened for two randomised clinical trials (RCTs) sponsored by AstraZeneca (AZ): SELECT-1 and SELECT-2 trials, but who do not meet eligibility criteria for those trials
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — Non interventional prospective data collection
  Other Names: Advanced second line patients

SUMMARY:
The recent development of therapies targeting specific biomarkers mutations is changing the standards of care and prognosis of patients with advanced NSCLC, but very few data are currently available on those emerging biomarkers. In addition, the correlation of biomarkers with patients' clinical outcomes in a standard of care setting is poorly understood. This study aims to address that need.

DETAILED DESCRIPTION:
The LUMINIST study will enrol patients who are ineligible for the SELECT-1 (NCT01933932) or SELECT-2 (NCT01750281)RCTs. Within this NIS patients will be followed longitudinally for treatment information and outcomes. The final dataset will enable linkage at the individual patient level of the clinical information datasets collected within LUMINIST to the exploratory biomarker data generated from samples collected as part of SELECT-1 screening. This will enable the examination of various molecular markers in patients with v-Ki-ras2 Kirsten Rat Sarcoma Viral Oncogene Homolog (KRAS) wild-type and some KRAS mutation positive (KRAS+) patients. The LUMINIST study aims to enable the investigation of various molecular segments in NSCLC, based on patient consent and where permitted by local legislation, some of which have not yet been discovered. The availability of a longitudinal dataset of clinical information linked to tumour samples will be a valuable tool to readily assess the clinical utility of potential new biomarkers. The determination of current standards of care and outcomes in future molecular segments of interest will provide valuable new insights to the scientific community.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent from the patient or next-of-kin for deceased patient at study entry, where this is mandated by local regulations
2. Female and male adults (according to each country regulations for age of majority)
3. Patients who are not eligible or choose not to enter selumetinib SELECT-1 or SELECT-2 trials
4. Patients with confirmed histological diagnosis of NSCLC

Exclusion Criteria:

1. Involved in the planning and/or conduct of this study (applies to both AZ staff and/or staff at the study site)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Advanced 2nd line NSCLC patients who are screened for two randomised clinical trials (RCTs) sponsored by AstraZeneca (AZ): SELECT-1 and SELECT-2 trials, but who do not meet eligibility criteria for those trials.
Sampling Method: Non-Probability Sample
Enrollment: 770 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 34 months
  The Overall Survival will be calculated from the first date of each line of therapy to end of follow-up or death, whichever occurs first.

SECONDARY OUTCOMES:
Progression Free survival (PFS) | Up to 34 months
  The length of time during and after the treatment of NSCLC that a patient lives with the disease but it does not progress (as defined by the Investigator).
Time to progression (TTP) | Up to 34 months
  The Time to Progression will be measured as the time from the first date of each line of therapy until the first date of documented disease progression. Time to Progression will be censored at the last tumour assessment available.
Duration of response (DOR) (complete or partial) | Up to 34 months
  The Duration of Response will be calculated as the time from the first documented complete response or partial response (whichever status is recorded first) until the first date of documented recurrence or progressive disease or death.
Complete response to treatment | Up to 34 months
  The complete response to treatment will be calculated as the percentage of patients per line of therapy having a complete response.
Healthcare resource utilisation (HRU) | Up to 34 months
  The number of hospitalisations, emergency room and outpatient visits, and the proportion of patients with a caregiver will be estimated.
Patients' characteristics | Up to 34 months
  The characteristics of the patients (Demographics (age, gender) smoking status, known mutations, tumour status and line of therapy) will be summarized descriptively by line of therapy.

OTHER OUTCOMES:
Overall Survival, Progression Free Survival, Time to Disease Progression, Duration of Response, Overall Response Rate and Healthcare Resource Utilisation | Up to 34 months
  The main outcomes will be stratified on biomarkers if interest and line of therapy
Prevalence of emerging biomarkers | Up to 34 months
  Prevalence of each biomarker will be calculated as the percentage of patients presenting a mutation/alteration/amplification
Treatment patterns among emerging biomarkers | Up to 34 months
  Treatments will be described by biomarkers to identify any emerging pattern.
Risk factors for non-response or resistance to standards of care | Up to 34 months
  Regression model will be used to estimate risk factors for non-response or resistance to standards of care, notably known and emerging biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Mariani, MD, Study Chair — AstraZeneca UK, MSD
Locations (85):
- Australia (4):
  - Research Site, Camperdown
  - Research Site, Darlinghurst
  - Research Site, Kurralta Park
  - Research Site, Wendouree
- Research Site, Salzburg, Austria
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Roeselare
- Bulgaria (2):
  - Research Site, Sofia
  - Research Site, Vratsa
- Canada (5):
  - Research Site, Edmonton
  - Research Site, Montreal
  - Research Site, Oshawa
  - Research Site, Regina
  - Research Site, Saskatoon
- Research Site, Santiago, Chile
- Research Site, Brest, France
- Germany (10):
  - Research Site, Bad Berka
  - Research Site, Cologne
  - Research Site, Großhansdorf
  - Research Site, Halle
  - Research Site, Homburg / Saar
  - Research Site, Löwenstein
  - Research Site, Moers
  - Research Site, München
  - Research Site, Ulm
  - Research Site, Würzburg
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Edelény
  - Research Site, Kaposvár
  - Research Site, Miskolc
- Israel (5):
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Kfar Saba
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (7):
  - Research Site, Bari
  - Research Site, Genova
  - Research Site, Livorno
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Parma
  - Research Site, Roma
- Research Site, Monterrey, Mexico
- Netherlands (3):
  - Research Site, 's-Hertogenbosch
  - Research Site, Amsterdam
  - Research Site, Bergen op Zoom
- Research Site, Lima, Peru
- Poland (5):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Sucha Beskidzka
  - Research Site, Szczecin
  - Research Site, Warsaw
- Portugal (5):
  - Research Site, Amadora-Lisbon
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Santa Maria da Feira
- Research Site, Cluj-Napoca, Romania
- Russia (4):
  - Research Site, Chelyabinsk
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Volgograd
- Spain (5):
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Vigo
  - Research Site, Zaragoza
- Sweden (2):
  - Research Site, Linköping
  - Research Site, Uppsala
- Turkey (Türkiye) (5):
  - Research Site, Ankara
  - Research Site, Erzurum
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Manisa
- Ukraine (7):
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kryvyi Rih, Dnipropetrovsk Region
  - Research Site, Kyiv
  - Research Site, Sumy
  - Research Site, Uzhhorod
- United Kingdom (4):
  - Research Site, Aberdeen
  - Research Site, Manchester
  - Research Site, Nottingham
  - Research Site, Wolverhampton

REFERENCES:
- See also: D1532R00004_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2997&filename=D1532R00004_CSR_Synopsis.pdf